CLINICAL TRIAL: NCT01911234
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Clinical Efficacy of Neovacs' TNF-Kinoid in Adult Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: Clinical Efficacy of TNF-Kinoid in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNF-K-006; 2013-001999-38 (EudraCT Number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — montanide ISA 51

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNF-Kinoid (Experimental): TNF Kinoid + ISA51
  Interventions: Biological: TNF-Kinoid
- Placebo (Placebo Comparator): Placebo + ISA51
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TNF-Kinoid — IM administration
  Other Names: ISA 51
  Arms: TNF-Kinoid
Other: Placebo — IM administration
  Other Names: ISA 51
  Arms: Placebo

SUMMARY:
The safety and immunogenicity of the TNF-Kinoid (TNF-K) have been evaluated in a phase II clinical study conducted in subjects with Rheumatoid arthritis. Preliminary results of clinical efficacy are promising.

The principal aim of the present study is to confirm the clinical efficacy of the TNF-K in subjects with Rheumatoid arthritis in whom treatment with methotrexate is not working anymore. Subjects who have never been treated with anti-TNFα monoclonal antibodies will be enrolled in this trial. In addition, the immune responses and the safety elicited by TNF-K will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has had a diagnosis of RA according to the revised ACR criteria (Aletaha et al. 2010) for at least 6 months.
* Has been treated with and tolerated MTX for at least 3 months prior to the first administration of study product, - Has at least four swollen joints/66 and/or four tender joints/68,
* Has CRP ≥ 10 mg/L at screening.
* Is positive for rheumatoid factor (RF) or anti-cyclic citrullinated peptides (CCP) antibodies at screening.

Exclusion Criteria:

* Has inflammatory rheumatic disease other than RA
* Has been treated with non-biological DMARDs/systemic immunosuppressives
* Has been treated with leflunomide within 12 weeks prior to first administration of study product.
* Has received intra-articular, intramuscular (IM), or intravenous (IV) corticosteroids
* Has received infliximab, etanercept, adalimumab, certolizumab, golimumab; another TNFα antagonist; or rituximab prior to the study.
* Has been treated with any other biological DMARDs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in DAS28-CRP between Month 6 and baseline. | Month 6

SECONDARY OUTCOMES:
Clinical responses defined as ACR20, ACR50, ACR70, SDAI, EULAR responses, changes in Tender and Swollen joint counts, DAS-28 and HAD-QI versus baseline | Several timepoints during 24 weeks study period
Immunogenicity: Anti-TNFα antibodies, Anti-TNFα neutralizing antibody activity, Anti-KLH antibodies by ELISA ; cytokines | Several timepoints during 24 weeks study period
Safety assessments will be conducted throughout the study and will include physical examinations, vital signs, clinical laboratory evaluations, and the recording of adverse events (AEs) | Several timepoints during 24 weeks study period

CONTACTS AND LOCATIONS:
Locations (31):
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- Georgia (4):
  - "Acad. V. Tsitlanadze Scientific-Practical Center of Rheumatology" LLC, Tbilisi
  - "Medi Club Georgia" LLC, Tbilisi
  - Diagnostic services LTD, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
- Hungary (3):
  - BKS Research Kft. Albert Schweitzer Kórhaz es Rendelőintezet-3. emelet, Hatvan
  - CRU Hungary Kft., Szikszó
  - Csolnoky Ferenc Kórház, Veszprém
- Lebanon (3):
  - Ain Wazein Hospital, Aïn Ouzaïn
  - University Medical Center Rizk Hospital, Beirut
  - Hammoud Hospital Univeristy Medical Center, Sidon
- IMSP Institutul de Cardiologie, Chisinau, Moldova
- University Clinic of Rheumatology, Skopje, North Macedonia
- Poland (3):
  - Osteomedic Sc, Bialystok
  - NZOZ "DOBRY LEKARZ" Specjalistyczne Poradnie Lekarskie, Krakow
  - Centrum Badań Klinicznych SC., Poznan
- Russia (4):
  - Municipal Clinical Hospital #4, Ivanovo
  - Regional Clinical Hospital for War Veterans, Kemerovo
  - City Clinical Hospital n.a.S.R.Mirotvortcev, Saratov
  - Clinical Hospital for Emergency Care n.a. N.V.Solovyev, Yaroslavl
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Institute for treatment and rehabilitation "Niska Banja"-Nis, Niška Banja
- Ukraine (9):
  - Donetsk City Clinical Hospital #5, Donetsk
  - Gusak Institute of Urgent and Recovery Surgery of AMSU, Donetsk
  - Municipal Health Care Institution "Kharkiv City Clinical Hospital #8", Kharkiv
  - Kyiv Out-patient hospital #2 of Shevchenko District, Kyiv
  - National medical academy of postgraduate education, Kiev regional clinical hospital, Kyiv
  - The Seventh Simferopol City Clinical Hospital, Simferopol
  - Municipal Institution "Central Hospital of Ordzhonikidze District", Zaporizhzhya
  - State Institution "Departmental Clinical Hospital of Railway Station Zaporizhzhya-2" of the State Enterprise "Prydniprovska Zaliznytsya", Zaporizhzhya
  - Zhitomir Regional Clinical Hospital named after O.F. Herbachevskogo, Zhytomyr